CLINICAL TRIAL: NCT01419704
Title: Phase I/II Pilot Study of Mixed Chimerism to Treat Hemoglobinopathies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study completed at site, no active participants.
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT-13881-012011
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Anemia, Sickle Cell; Complex and Transfusion-dependent Hemoglobinopathies; Thalassemia; Diamond-Blackfan Anemia; Bone Marrow Failure Syndromes; Alpha-Thalassemia; Beta-Thalassemia
Keywords: other hemoglobinopathies; chimerism; sickle cell; thalassemia; Marrow/Enriched Hematopoetic Stem Cell Transplant
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Anemia, Diamond-Blackfan; Bone Marrow Failure Disorders; alpha-Thalassemia; beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hemoglobinopathies diagnosed patients (Experimental): Recipients diagnosed with Hemoglobinopathies are treated with an enriched hematopoetic stem cell infusion from living donor bone marrow
  Interventions: Biological: Enriched Hematopoetic Stem Cell Infusion

INTERVENTIONS:
Biological: Enriched Hematopoetic Stem Cell Infusion — Enriched Hematopoetic Stem Cell Infusion

SUMMARY:
The goal of this research study is to establish chimerism and avoid graft-versus-host disease in patients with hemoglobinopathies.

DETAILED DESCRIPTION:
This proposal is a phase I/II feasibility study to demonstrate that mixed chimerism can be established with minimal risk in recipients with hemoglobinopathies treated with Campath-1H-based nonmyeloablative conditioning and graft engineering to reduce the risk of Graft Versus Host Disease (GVHD), but preserve engraftment of donor cells.

ELIGIBILITY:
1. Inclusion Criteria

   The following criteria are established to identify subjects with hemoglobinopathies, hematologic or bone marrow failure syndromes who have a high predicted morbidity and are at risk for early mortality:
   * Patients with alpha or beta thalassemia major.
   * Patients with Diamond-Blackfan anemia and other bone marrow failure syndromes, characterized by severe chronic anemia.
   * Patients with other complex and transfusion-dependent hemoglobinopathies, including sickle cell disease.
   * Patients with sickle disease who have one or more of the following:

     * Overt or silent stroke
     * Neurocognitive impairment
     * Pain crises 2 or more episodes per year for past year
     * One or more episodes of acute chest syndrome
     * Osteonecrosis involving 1 or more joints
     * Evidence of retinopathy
     * Priapism
     * Microalbuminuria or evidence of sickle cell nephropathy
     * Alloimmunization

   Subjects must also meet all of the following general inclusion criteria:
   * Subjects must have a related donor which can consist of Histocompatibility Leukocyte Antigen (HLA)-matched donor up to haploidentical match, mismatched for 1, 2 or 3 HLA-A, B or -DR loci.
   * Subjects must have adequate cardiopulmonary function as documented by echocardiogram or radionuclide scan. (Shortening fraction >26% or ejection fraction >40% or ≥ 80% of normal value for age).
   * Subjects must have adequate pulmonary function documented by Forced expiratory volume in 1 second (FEV1) of ≥ 50% of predicted for age and/or Diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) ≥50% of predicted for age for patients > 10 years of age.
   * Subjects must have adequate hepatic function as demonstrated by a serum albumin ≥ 3.0 mg/dL, and serum glutamic pyruvic transaminase (SGPT) or serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 5 times the upper limit of normal. Liver biopsy or a liver MRI is necessary if the patient has received chronic transfusions for over a year and/or has a ferritin level of ≥ 1600.
   * Subjects must have adequate renal function as demonstrated by a serum creatinine less than or equal to 2 mg/dL. If serum creatinine is ≥ 2 mg/dL, then a creatinine clearance test or nuclear medicine GFR should document GFR of ≥ 50 ml/min/1.73 m2.
   * Subjects or legal guardians must give written informed consent.
   * Female patients of childbearing potential cannot be pregnant or lactating/breast-feeding and must be either surgically sterile, postmenopausal (no menses for the previous 12 months), or must be practicing an effective method of birth control as determined by the investigator (e.g., oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy).
   * Less than or equal to 45 years of age.
2. Exclusion Criteria

   * Patients with cirrhosis, extensive bridging hepatic fibrosis, or active hepatitis are excluded from enrollment.
   * Uncontrolled infection or severe concomitant diseases, which in the judgment of the Principal Investigator, indicate that the patient could not tolerate reduced intensity transplantation.
   * Severe impairment of functional performance as evidenced by a Karnofsky score <70% (patients ≥16 years old) or Lansky (children <16 years old) score <70%
   * Renal insufficiency (GFR <50 ml/min/1.73 m2).
   * Subjects with a positive human immunodeficiency virus (HIV) antibody test result.
   * Subjects who are pregnant, as indicated by a positive serum human chorionic gonadotrophin (HCG) test.
   * Subjects whose only donor is pregnant at the time of intended transplant.
   * Subjects of childbearing potential who are not practicing adequate contraception as defined by the investigator at the site.
   * Allogeneic hematopoietic stem cell transplant within the previous 1 year.
   * Subjects must not have had previous radiation therapy that would preclude total body irradiation (TBI) (as determined by a radiation therapist).
   * Jehovah's Witness unwilling to be transfused .
   * Uncontrolled hypersplenism.
   * Severe alloimmunization with inability to guarantee a supply of adequate packed red blood cell (PRBC) donors.
   * Subjects with thalassemia who are Lucarelli Class 3
   * Fanconi anemia.
   * Insufficient funds for the bone marrow processing costs

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Proportion of Hemoglobin A and S | one month to three years
  Red blood cell contents by hemoglobin electrophoresis

SECONDARY OUTCOMES:
Enriched Hematopoetic Stem Cell Engraftment | One month to three years

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, MD, Study Director — Talaris Therapeutics Inc.
Locations (3):
- United States (3):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided